CLINICAL TRIAL: NCT02480972
Title: Hepatic Fibrosis Assessment Using Multiparametric Magnetic Resonance Imaging (MRI)
Brief Title: Hepatic Fibrosis Assessment Using Multiparametric Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-082-618
Record Dates: First submitted 2015-06-18; First posted 2015-06-25 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Fibrosis; Cirrhosis
Keywords: fibrosis; cirrhosis; MRI
MeSH Terms: conditions — Fibrosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic resonance imaging (Other): multiparametric MRI including perfusion, diffusion, MR fat quantification and MR elastography
  Interventions: Procedure: magnetic resonance imaging

INTERVENTIONS:
Procedure: magnetic resonance imaging — multiparametric MRI as follows:
  1. diffusion weighted imaging using multiple b-values
  2. Fat quantification sequence
  3. perfusion MRI using ECCM agent
  4. MR elastography
     ------------------------------------
  5. routine MRI using hepatocyte specific agent (optional in patients with focal liver lesion)
  Other Names: MRI

SUMMARY:
The purpose of this study is to assess degree of hepatic fibrosis using multiparametric MRI for investigating difference between normal or early fibrosis and advanced fibrosis.

DETAILED DESCRIPTION:
In patients with liver parenchymal disease or normal liver parenchyma who are scheduled to undergo either liver resection or liver biopsy are included.

Referred patients undergo multiparametric MRI including perfusion, diffusion, elastography and fat quantification before surgery or biopsy.

The pathophysiologic changes are evaluated using multiparametric MRI, and compared between normal/early fibrosis and advanced fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo liver resection for focal liver lesion
* patients who are scheduled to undergo liver resection or percutaneous biopsy for diffuse parenchymal disease
* liver donor candidate who are scheduled to undergo preoperative liver biopsy or liver resection
* AND patients/living donor candidates who sign informed consent

Exclusion Criteria: Patients who have at least one of followings are excluded.

* Patients who are contraindication for MRI contrast enhanced MRI.
* Premenopausal female patients who are pregnant.
* Patients who are physically compromised to acquire liver MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
difference of portal flow between no or early hepatic fibrosis and advanced hepatic fibrosis | in three years

SECONDARY OUTCOMES:
difference of arterial flow between no or early hepatic fibrosis and advanced hepatic fibrosis | in three years
difference of liver stiffness value between no or early hepatic fibrosis and advanced fibrosis | in three years
monitoring of transient dyspnea after contrast media injection | in three years

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No